CLINICAL TRIAL: NCT01979341
Title: Dual Trigger With Gonadotropin-releasing Hormone Agonist (GnRHa) and Human Chorionic Gonadotropin (hCG) to Optimize ICSI Reproductive Outcomes
Brief Title: The Effect of a Dual Trigger on Intracytoplasmic Sperm Injection (ICSI) Reproductive Outcomes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: treatment strategy changed
Sponsor: Antalya IVF (Other)
Responsible Party: Principal Investigator, Kevin Coetzee, Scientific Advisor, Antalya IVF
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AntalyaIVF-RCT-dual trigger; App. No. 01042013/103 (Other: Turkish Health Ministry Ethics Committee/Akdeniz University Ethics Committee)
Record Dates: First submitted 2013-11-01; First posted 2013-11-08 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-05

CONDITIONS: Pregnancy; Ovarian Hyperstimulation Syndrome
Keywords: dual trigger; hCG; GnRH agonist; ICSI; pregnancy; OHSS
MeSH Terms: conditions — Ovarian Hyperstimulation Syndrome | interventions — Chorionic Gonadotropin; Triptorelin Pamoate; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dual trigger (Active Comparator): final oocyte maturation trigger using 6500 IU Ovitrelle (hCG) plus 0.2mg triptorelin acetate (GnRH agonist)
  Interventions: Procedure: final oocyte maturation trigger
- hCG trigger (Active Comparator): final oocyte maturation trigger using 6500 IU Ovitrelle (hCG)
  Interventions: Procedure: final oocyte maturation trigger
- agonist trigger (Active Comparator): final oocyte maturation trigger using 0.2mg triptorelin acetate (GnRH agonist)
  Interventions: Procedure: final oocyte maturation trigger

INTERVENTIONS:
Procedure: final oocyte maturation trigger — when ≥3 follicles reach 17mm patients will be randomized to receive one of two types of trigger for final oocyte maturation; dual trigger: GnRH agonist plus hCG (both full doses) hCG only: full dose of hCG only
  Other Names: dual trigger: 6500 IU Ovitrelle (hCG) plus 0.2mg triptorelin acetate (GnRH agonist); hCG trigger: 6500 IU Ovitrelle (hCG); agonist trigger: 0.2mg triptorelin acetate (GnRH agonist)

SUMMARY:
The use of antagonist controlled ovarian stimulation protocols has allowed the use of GnRH agonist to be used for final oocyte maturation. The use of GnRH agonist as ovulation trigger has been shown to reduce the risks for ovarian hyperstimulation syndrome (OHSS), but its sole use results in reduced embryo implantation due to luteal phase insufficiency. The combination of GnRH agonist and variable doses of hCG for final oocyte maturation has been shown to overcome the luteal phase insufficiency effecting endometrial receptivity.

In this study the investigators will test the hypothesis that using GnRH agonist (0.2mg Triptorelin) and a full dose of hCG (6500IU Ovitrelle) for final oocyte maturation in normoresponders will increase oocyte maturity, embryo quality and embryo implantation and reduce ovarian hyperstimulation syndrome, as compared to the traditional hCG (full dose) alone trigger.

ELIGIBILITY:
Inclusion Criteria:

* Age; < 40 years
* Cycle number; cycles 1 or 2
* Antral follicle count; >10 and <25
* BMI; >18 and <30
* Normogonadotrophic cycle length; 24 to 25 days
* Male; ejaculated semen only

Exclusion Criteria:

* Presence of endocrine disorders; (diabetes mellitus, hyperprolactinemia, thyroid dysfunction, congenital adrenal hyperplasia, Cushing syndrome, or polycystic ovary syndrome)
* Previous major uterine surgery (that would affect endometrial receptivity)

Secondary exclusion criteria

* <5 follicles at the time of trigger
* <2 full formed blastocyst on day 5 of embryo culture

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2016-06 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
embryo implantation rate | 12 months
  the number of fetal sacs per embryo transferred to a patient's uterus

SECONDARY OUTCOMES:
oocyte maturation | 12 months
  the percentage of oocytes that are at the metaphase II (nuclear mature) stage at the time of oocyte collection
Ovarian hyperstimulation syndrome | 12 months
  a complication arising from ovarian hyperstimulation with the use of exogenous hormones and ovulation induction

OTHER OUTCOMES:
clinical pregnancy | 12 months
  the number of patients with an ultrasound confirmed fetal heart 7 weeks after the transfer of embryos to patient uteruses

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Bulut, MD, Principal Investigator — Antalya IVF; Kemal Ozgur, MD, Principal Investigator — Antalya IVF
Locations (1):
- Antalya IVF, Antalya, Antalya, Turkey (Türkiye)